CLINICAL TRIAL: NCT04704401
Title: Collection of Long-Term Follow-up Medical Events in Patients Included in the Meta-analysis "Sleep Apnea Syndrome and Arterial Stiffness"
Brief Title: Long-Term Follow-up in Patients Included in the Meta-analysis "Sleep Apnea Syndrome and Arterial Stiffness"
Acronym: PWV follow-up
Status: Terminated | Type: Observational
Why Stopped: recruitment difficulty
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC20.373; 2020-A03065-34 (Other: ID RCB)
Record Dates: First submitted 2020-12-07; First posted 2021-01-11 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Sleep Apnea
Keywords: Sleep apnea; Follow-up; Cardiovascular event; Metabolic event; incident cancer; Death
MeSH Terms: conditions — Sleep Apnea Syndromes; Death | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients PWV follow-up: Patients included in the meta-analysis "sleep apnea syndrome and arterial stiffness" and contacted by phone for the collection of cardiovascular and metabolic events, incident cancers and deaths, through a structured questionnaire.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Structured questionnaire to collect cardiovascular and metabolic events, incident cancers and deaths that have occured, as weel as information on CPAP, through telephone interview.

SUMMARY:
The meta-analysis "sleep apnea syndrome and arterial stiffness" includes data from 893 patients initially included in 9 studies conducted by the EFCR Department of the CHUGA between 2006 and 2015, presenting a sleep apnea syndrome (SAS) with exploration of their arterial stiffness via the measurement of pulse wave velocity (PWV).

Currently, we do not have long-term follow-up data for these patients.

The first objective of the "PWV Follow-up" project is to collect cardiovascular events in these patients through telephone interviews and a structured questionnaire to determine the prevalence of these events. The prevalence of metabolic events, incident cancers and deaths will be also determined as secondary objectives through the same questionnaire.

Others secondary objectives are to evaluate the impact of continuous positive airway pressure (CPAP, the reference treatment for OSA) on the occurrence of cardiovascular and metabolic events and incident cancers, as this is still discussed in the literature.

DETAILED DESCRIPTION:
The meta-analysis "sleep apnea syndrome and arterial stiffness" includes data from 893 patients initially included in 9 studies conducted by the EFCR Department of the CHUGA between 2006 and 2015, presenting a sleep apnea syndrome (SAS) with exploration of their arterial stiffness via the measurement of pulse wave velocity (PWV).

The 9 studies were referred as : ADISAS (NCT011968), AGIRSASADOM (NCT010902), BPCO (NCT004044), BPCO-SAS (NCT01195064), DIAMETASAS, Aortic Dissection (NCT01068691), INFRASAS (NCT010892), VALSAS (NCT004094), NIV-OHS (NCT006030).

The objective of this meta-analysis on individual data was to understand the relationship between the severity of the sleep apnea syndrome (measured by the apnea + hypopnea index) and arterial rigidity at the time of diagnosis of SAS.

Currently, we do not have long-term follow-up data for these patients.

The first objective of the "PWV Follow-up" project is to collect cardiovascular events in these patients through telephone interviews and a structured questionnaire to determine the prevalence of these events. The prevalence of metabolic events, incident cancers and deaths will be also determined as secondary objectives through the same questionnaire.

Others secondary objectives are to evaluate the impact of continuous positive airway pressure (CPAP, the reference treatment for OSA) on the occurrence of cardiovascular and metabolic events and incident cancers, as this is still discussed in the literature.

ELIGIBILITY:
Inclusion Criteria:

* already included in the meta-analysis "sleep apnea syndrome and arterial stiffness".

Exclusion Criteria:

* refusal to participate
* family not reachable and death not identified in the Hospital medical base
* persons under judicial protection (article L1122-2 of the Public Health Code) and patients under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sleep apnea patients included in the meta-analysis "sleep apnea syndrome and arterial stiffness"
Sampling Method: Non-Probability Sample
Enrollment: 321 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-08-29 (Actual)

PRIMARY OUTCOMES:
Prevalence of cardiovascular events | up to 15 years
  Prevalence of cardiovascular events during the follow-up of patients included in the meta-analysis "sleep apnea syndrome and arterial stiffness", through a structured questionnaire.

SECONDARY OUTCOMES:
Prevalence of metabolic events | up to 15 years
  Prevalence of metabolic events during the follow-up of patients included in the meta-analysis "sleep apnea syndrome and arterial stiffness", through a structured questionnaire.
Prevalence of incident cancers | up to 15 years
  Prevalence of incident cancers during the follow-up of patients included in the meta-analysis "sleep apnea syndrome and arterial stiffness", through a structured questionnaire..
Prevalence of deaths | up to 15 years
  Prevalence of deaths during the follow-up of patients included in the meta-analysis "sleep apnea syndrome and arterial stiffness", through a structured questionnaire.
Effect of CPAP treatment on the cardiovascular events occurrence | during 6 months
  Mean CPAP observance (h/night) of patients included in the meta-analysis "sleep apnea syndrome and arterial stiffness" to determine its impact on the cardiovascular events occurrence.
Effect of CPAP treatment on the metabolic events occurrence | during 6 months
  Mean CPAP observance (h/night) of patients included in the meta-analysis "sleep apnea syndrome and arterial stiffness" to determine its impact on the metabolic events occurrence.
Effect of CPAP treatment on the incident cancers occurrence | during 6 months
  Mean CPAP observance (h/night) of patients included in the meta-analysis "sleep apnea syndrome and arterial stiffness" to determine its impact on the incident cancers occurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis PEPIN, MD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bironneau V, Tamisier R, Trzepizur W, Andriantsitohaina R, Berger M, Goupil F, Joyeux-Faure M, Jullian-Desayes I, Launois S, Le Vaillant M, Martinez MC, Roche F, Pepin JL, Gagnadoux F. Sleep apnoea and endothelial dysfunction: An individual patient data meta-analysis. Sleep Med Rev. 2020 Aug;52:101309. doi: 10.1016/j.smrv.2020.101309. Epub 2020 Mar 13. PMID 32234658